CLINICAL TRIAL: NCT02852382
Title: The Effects of Scalp Block on Haemodynamic Response and Postoperative Pain in
Brief Title: The Effects of Scalp Block on Haemodynamic Response and Postoperative Pain in Posterior Fossa Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Eren Fatma Akcil, Staff anesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cerrahpasa Neuro
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Posterior Fossa Tumors
Keywords: scalp block; local infiltration
MeSH Terms: conditions — Infratentorial Neoplasms | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- scalp block (Active Comparator): In this arm, after general anesthesia, before surgery and head pin placement, scalp block will be applied. Scalp block will be performed with bupivacaine (Marcaine 5 mg/mL, 0,5% bupivacaine); nervus supraorbitalis, nervus supratrochlearis, n. auriculotemporalis, nervus zygomaticotemporalis, nervus occipitalis majoris and minoris will be bilaterally blocked with 2-3 ml bupivacaine.
  Interventions: Drug: Bupivacaine; Drug: morphine patient controlled analgesia
- local infiltration (Active Comparator): In this arm, after general anesthesia, before surgery, 20 ml 0,5% bupivacaine (Marcaine 5 mg/ml, 0,5% bupivacaine) will be infiltrated to head pin points and skin incision area.
  Interventions: Drug: Bupivacaine; Drug: morphine patient controlled analgesia
- control (Placebo Comparator): In this arm, neither scalp block, nor local infiltration will be performed.
  Interventions: Drug: morphine patient controlled analgesia

INTERVENTIONS:
Drug: Bupivacaine — In the scalp block and local infiltration arms; bupivacaine %0,5 will be used.
  Other Names: Marcaine
  Arms: local infiltration; scalp block
Drug: morphine patient controlled analgesia — End of the surgery all of the patients in 3 groups will receive morphine patient controlled analgesia (PCA) including 1mg/ml morphine. The PCA was set to administer a bolus dose of 1 mg on demand with a lockout period of 10 minutes and maximum 25 mg for 4 hours.
  Other Names: MORPHİNE PCA

SUMMARY:
This study evaluate the effects of scalp block versus local infiltration on haemodynamic response to head pin replacement and skin incision and postoperative analgesia in posterior fossa surgery

DETAILED DESCRIPTION:
In this study 15 patients will receive scalp block with bupivacaine, 15 patients will receive local infiltration with bupivacaine and 15 patients will receive placebo before surgery. The haemodynamic response to head pin replacement and skin incision will be recorded. Postoperatively all patients will have a patient controlled analgesia (PCA) device containing morphine (1 mg/ml) for analgesia. Visual analogue scale (VAS) for pain evaluation, sedation scores, and also postoperative morphine consumption will be evaluated and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Posterior fossa surgery
* Preoperative GlasGow Coma Score: 15/15

Exclusion Criteria:

* Allergy to bupivacaine
* Uncontrolled hypertension
* Coagulopathy
* Cerebrovascular disease
* Earlier craniotomy

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Heart rate response to head pin replacement and skin incision | Intraoperative
  heart rates (beats per minute) will be recorded before induction, before block, before head pinning, head pinning, head pin 5. and 10. minutes, skin incision
Systolic arterial pressure response to head pin replacement and skin incision | Intraoperative
  Systolic arterial pressures (mmHg) will be recorded in before induction, before block, before head pinning, head pinning, head pin 5. and 10. minutes, skin incision
Diastolic arterial pressure response to head pin replacement and skin incision | Intraoperative
  Diastolic arterial pressures (mmHg) will be recorded before induction, before block, before head pinning, head pinning, head pin 5. and 10. minutes, skin incision
mean arterial pressure response to head pin replacement and skin incision | Intraoperative
  Mean arterial pressures (mmHg) will be recorded in will be recorded before induction, before block, before head pinning, head pinning, head pin 5. and 10. minutes, skin incision

SECONDARY OUTCOMES:
postoperative pain | 30. minute, 1.,2.,6.,12.,24. hours pain scores (visual analogue score=VAS)
  pain scores (visual analogue score=VAS) will be evaluated.
morphine consumption | 30. minute, 1.,2.,6.,12.,24. hours
  morphine dosage used (mg) will be recorded in this time periods

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Tunali, Professor, Study Director — Istanbul University Cerrahpasa Medical Faculty Department Anesthesiology and Reanimation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Geze S, Yilmaz AA, Tuzuner F. The effect of scalp block and local infiltration on the haemodynamic and stress response to skull-pin placement for craniotomy. Eur J Anaesthesiol. 2009 Apr;26(4):298-303. doi: 10.1097/EJA.0b013e32831aedb2. PMID 19262392
- [Result] Hansen MS, Brennum J, Moltke FB, Dahl JB. Pain treatment after craniotomy: where is the (procedure-specific) evidence? A qualitative systematic review. Eur J Anaesthesiol. 2011 Dec;28(12):821-9. doi: 10.1097/EJA.0b013e32834a0255. PMID 21971206
- [Result] Verchere E, Grenier B, Mesli A, Siao D, Sesay M, Maurette P. Postoperative pain management after supratentorial craniotomy. J Neurosurg Anesthesiol. 2002 Apr;14(2):96-101. doi: 10.1097/00008506-200204000-00002. PMID 11907388
- [Result] Jellish WS, Leonetti JP, Sawicki K, Anderson D, Origitano TC. Morphine/ondansetron PCA for postoperative pain, nausea, and vomiting after skull base surgery. Otolaryngol Head Neck Surg. 2006 Aug;135(2):175-81. doi: 10.1016/j.otohns.2006.02.027. PMID 16890064
- [Result] Irefin SA, Schubert A, Bloomfield EL, DeBoer GE, Mascha EJ, Ebrahim ZY. The effect of craniotomy location on postoperative pain and nausea. J Anesth. 2003;17(4):227-31. doi: 10.1007/s00540-003-0182-8. PMID 14625709
- [Result] Schessel DA, Nedzelski JM, Rowed D, Feghali JG. Pain after surgery for acoustic neuroma. Otolaryngol Head Neck Surg. 1992 Sep;107(3):424-9. doi: 10.1177/019459989210700314. PMID 1408229